CLINICAL TRIAL: NCT03646695
Title: ILM Flap Transposition Versus ILM Peeling for Macular Holes: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department of Ophthalmology, Professor, Principal Investigator, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILM flap
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILM flap (Experimental): vitrectomy with ILM flap transposition and gas-tamponade will be performed
  Interventions: Procedure: ILM flap transposition
- ILM peeling (Active Comparator): vitrectomy with ILM peeling and gas-tamponade will be performed
  Interventions: Procedure: ILM peeling

INTERVENTIONS:
Procedure: ILM flap transposition — during ILM flap Transposition, an ILM flap is placed on the macular hole
  Arms: ILM flap
Procedure: ILM peeling — during ILM Peeling the ILM is removed around the macular hole
  Arms: ILM peeling

SUMMARY:
Patients with macular hole <400µm will be randomized for ILM flap Transposition and ILM Peeling for surgical repair of macular holes

DETAILED DESCRIPTION:
Patients with macular hole with a diameter larger than 400µm have better sucess with ILM flap transposition, but there are no data published examining the outcome of macular hole with a diameter <400µm. Therefore, patients with macular hole with a diameter <400µm will be randomized for ILM flap transposition and ILM peeling for surgical repair of macular holes

ELIGIBILITY:
Inclusion Criteria:

* macular hole with a diameter <400µm

Exclusion Criteria:

* Prior ILM peeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
closure of the macular hole | 3 months
  closure of the macular hole will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Professor, Principal Investigator — Head of Department of Ophthalmology, Professor, Principal Investigator
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Austria